CLINICAL TRIAL: NCT03107910
Title: Novel Stigma/Structural Interventions for HIV/STI Testing
Brief Title: Stigma and Online Counseling to Increase HIV/STI Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Eaton, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: H16-087; R01MH109409 (NIH)
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: HIV/STI Testing

STUDY DESIGN:
Intervention Model Description: This project is 2 x 2 factorial approach designed to test an intervention that is aimed at increasing HIV/STI testing uptake among BMSM; this approach includes testing HIV/STI stigma focused counseling, and online HIV/STI test counseling with at-home, self-administered HIV and STI test kits.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator are masked to study intervention assignment. Participants are informed that they are randomly assigned to conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Stigma Counseling (Other): Single session, stigma focused, anticipated HIV stigma counseling will be provided. Intervention will include a focus on barriers to testing.
  Interventions: Behavioral: Stigma and Structural Interventions; Behavioral: Health Information Seeking
- Control Health Information (Other): Single session, online health information seeking and evaluation. HIV/STI testing appointments are provided online. Stigma and Structural Interventions
  Interventions: Behavioral: Stigma and Structural Interventions; Behavioral: Health Information Seeking

INTERVENTIONS:
Behavioral: Stigma and Structural Interventions — Stigma focused counseling to address HIV anticipated stigma and online video chatting for HIV/STI testing will be assessed. Stigma and Structural Interventions
Behavioral: Health Information Seeking — Seeking and evaluating online health information will be assessed.

SUMMARY:
The alarmingly high rates of HIV/STI (sexually transmitted infections) observed among Black men who have sex with men (BMSM) necessitate a new model for engaging BMSM. New approaches include addressing stigma related concerns and structural barriers in order to increase HIV/STI testing uptake. This research includes a 2 x 2 factorial design to test an intervention that is aimed at increasing HIV/STI testing uptake among BMSM; this design includes testing HIV/STI stigma focused counseling, and online HIV/STI test counseling with at-home, self-administered HIV and STI test kits.

DETAILED DESCRIPTION:
This research is aimed at conducting structural and stigma-focused interventions to increase HIV and STI testing uptake among Black men who have sex with men (BMSM). The research is focused on this population due to the alarmingly high rates of HIV/STI (sexually transmitted infections) among BMSM- this group has experienced elevated rates of HIV incidence and prevalence since the beginning of the US epidemic, and current estimates demonstrate that although BMSM make up only 0.2% of the population they make up 22% of new HIV infections. The investigator have documented a 5.1% annual HIV incidence and a 35% HIV prevalence among BMSM. Health care models are failing to engage BMSM at all points of the HIV care continuum including the seek and test components. The CDC recommends that individuals at substantial risk for HIV be tested for HIV/STI every three to six months; however, this goal is not being achieved and, therefore, a new approach to engaging BMSM is needed. To address these shortcomings and based on preliminary studies, the investigators are conducting a 2 x 2 factorial design study to evaluate a model that is aimed at increasing HIV/STI testing uptake among BMSM. The investigators will test a stigma-focused intervention as stigma is a known deterrent to HIV/STI testing, yet little has been done to address this factor; and, the investigators will evaluate HIV/STI test counseling delivered online (in conjunction with at-home HIV/STI test kits) as this delivery of testing may remove key barriers to reaching BMSM in need of HIV/STI related care services. Specific Aim 1: Assess HIV/STI testing uptake at scheduled HIV/STI test counseling appointments during the 12 month follow-up period. 500 BMSM will be randomly assigned to one of four conditions: (a) receive CDC-based risk reduction counseling and scheduled for in-office HIV/STI test counseling appointments, (b) receive HIV stigma-enhanced intervention and scheduled for in-office HIV/STI test counseling appointments, (c) receive CDC-based risk reduction counseling and scheduled for online, via video calling, HIV/STI test counseling appointments, or (d) receive HIV stigma-enhanced intervention and scheduled for online, via video calling, HIV/STI test counseling appointments. Specific Aim 2: Evaluate mediating (key theoretical stigma variables) factors collected via assessments at 3, 6, and 12 month follow-ups. Specific Aim 3: Conduct an economic evaluation to determine the costs of the office-based and online-based HIV/STI test delivery formats from both a community-based payer perspective and a comprehensive societal perspective that includes all costs. This project has the potential to exert a sustained and powerful impact not only on approaches to engaging BMSM, but to improving HIV/STI testing uptake which will likely improve multiple health outcomes among BMSM. If effective, this approach to improving HIV/STI testing uptake would be available for dissemination immediately and would fit within resource limited settings such as community based organizations and health departments.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* Transgender women who have sex with men
* 18 years of age and older
* Reside in Atlanta metro area.
* Other criteria may apply

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males, transgender women
Enrollment: 500 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
HIV/STI testing uptake | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Eaton, PhD, Principal Investigator — SHARE Project
Locations (1):
- SHARE Project, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Eaton LA, Huedo-Medina T, Earnshaw VA, Kalichman M, Watson RJ, Driver R, Chandler CJ, Kalinowski J, Kalichman SC. Randomized Clinical Trial of Stigma Counseling and HIV Testing Access Interventions to Increase HIV Testing Among Black Sexual Minority Men and Transwomen. Prev Sci. 2024 May;25(4):650-660. doi: 10.1007/s11121-023-01603-4. Epub 2023 Oct 29. PMID 37898978